CLINICAL TRIAL: NCT00378014
Title: Presentation of Renal Function in Liver Transplant Recipients With Certican Therapy: PROTECT Study A Twelve-month, Multicenter, Randomized, Open-label Study of Safety, Tolerability and Efficacy of Certican-based Regimen Versus Calcineurin Inhibitor-based Regimen in de Novo Liver Transplant Recipients
Brief Title: Preservation of Renal Function in Liver Transplant Recipients With Certican Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001HDE10; 2005-002920-32
Record Dates: First submitted 2006-09-15; First posted 2006-09-19 (Estimated); Results first posted 2014-07-03 (Estimated); Last update posted 2015-02-06 (Estimated); Status verified 2015-01

CONDITIONS: Liver Transplantation
Keywords: Liver transplantation, everolimus, CNI
MeSH Terms: interventions — Everolimus; Basiliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Everolimus (Experimental): Basiliximab plus everolimus-based immunosuppressive regimen following the reduction and cessation of initial CNI regimen plus optional steroids according to local best practice
  Interventions: Drug: basiliximab; Drug: CNI
- Calcineurin Inhibitor (CNI) (Active Comparator): Basiliximab plus CNI-based immunosuppressive regimen according to local best practice plus optional steroids according to local best practice
  Interventions: Drug: everolimus; Drug: basiliximab; Drug: CNI

INTERVENTIONS:
Drug: everolimus — Start dose of everolimus was 1.5 mg in the morning followed by 1.5 mg in the evening. After one week, the dose was adjusted to achieve trough levels between 5-12 ng/mL. Once trough levels were above 5ng/mL, the CNI dose was reduced to 70%. At week 8 post-baseline (latest at week 16 post baseline), CNI was completely discontinued. For patients receiving Ciclosporin A (CiA) as CNI, the everolimus dosage was adjusted to achieve a trough level of 8-12 ng/mL, prior to discontinuation of CiA. After discontinuation of CNI, everolimus was maintained at a trough level of 5-12 ng/mL.
  Other Names: certican
  Arms: Calcineurin Inhibitor (CNI)
Drug: basiliximab — All patients who met the eligibility criteria were treated with 2 doses of basiliximab on Day 0 (transplantation) and Day 4.
  Other Names: simulect
Drug: CNI — Patients who met the screening eligibility received CNI-based immunosuppressive therapy for 1 month. Then at week 4 (or week 8 at maximum), patients randomized to the CNI arm continued on CNI-based immunosuppressive therapy.

SUMMARY:
The study is designed to show that everolimus initiation together with reduction and thereafter discontinuation of calcineurin inhibitor (CNI) will improve significantly renal function in de novo liver transplant recipients as compared to continuation of CNI-based treatment.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 18 - 70 years old
* Liver transplant recipient (living or deceased donor)
* Patients in whom an allograft biopsy will not be contraindicated

Exclusion Criteria:

* Recipients of multiple solid organ transplants or patients that have already received a transplant in the past
* HCV positive patients who need an active anti-viral treatment (HCV- positive patients without active antiviral treatment are allowed)
* HIV positive patients
* Patients who are breast feeding
* Patients with a current severe systemic infection
* Presence of any hypersensitivity to drugs similar to Certican® (e.g. macrolides)
* Preexisting (i.e. not related to CNI-damage) renal dysfunction that, according to the judgment of the investigator, will not significantly improve after transplantation (i.e., for example, patients that are expected to have a cGFR below 50ml/min at 4 weeks post transplantation)
* Patients that have received Simulect prior to this study.
* Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2006-08; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (16):
- Austria (2):
  - Novartis Investigative Site, Innsbruck
  - Novartis Investigative Site, Vienna
- Germany (10):
  - Novartis Investigative Site, Berlin, Germany
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Regensburg
  - Novartis Investigative Site, Tübingen
- Netherlands (2):
  - Novartis Investigative Site, Groningen
  - Novartis Investigative Site, Rotterdam
- Switzerland (2):
  - Novartis Investigative Site, Zurich, Switzerland
  - Novartis Investigative Site, Geneva

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The core study consisted of 2 periods: 1) during the first one-month period, 276 eligible participants received the same CNI-based immunosuppressive therapy prior to randomization; 2) during the second 11-month study period, 203 participants eligible participants were randomized in a 1:1 ratio to one of the two treatment arms.
Period: Core (Randomization to Month 11)
Arm/Group | Everolimus | Calcineurin Inhibitor (CNI)
Started | 101 | 102
Intent-to-treat (ITT) Population | 96 (ITT contained all randomized patients who had at least one post baseline GFR measurement.) | 98 (ITT contained all randomized patients who had at least one post baseline GFR measurement.)
Completed | 87 | 90
Not Completed | 14 | 12
Not completed — Adverse Event | 1 | 0
Not completed — Graft loss | 1 | 2
Not completed — Death | 5 | 3
Not completed — Administrative Problems | 2 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 5 | 2
Not completed — Protocol deviation | 0 | 1
Not completed — Lack of Efficacy | 0 | 1
Period: Extension (Month 12 to Month 59)
Arm/Group | Everolimus | Calcineurin Inhibitor (CNI)
Started | 41 | 40
Completed | 27 | 26
Not Completed | 14 | 14
Not completed — Adverse Event | 8 | 7
Not completed — Death | 1 | 2
Not completed — Administrative problems | 1 | 0
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Lack of Efficacy | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Everolimus | Calcineurin Inhibitor (CNI) | Total
Number analyzed (Participants) | 96 | 98 | 194
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.3 (9.9) | 52.9 (10.1) | 52.6 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 30 | 72
  Male | 54 | 68 | 122

OUTCOME MEASURES:

1. Primary Outcome: Calculated Glomerular Filtration Rate (cGFR)
Description: This outcome measure evaluated renal function by assessing the calculated GFR based on the Cockcroft-Gault formula.
Time Frame: Month 11
Population: ITT
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Everolimus | Calcineurin Inhibitor (CNI)
Number analyzed (Participants) | 96 | 98
mL/min | 87.9 (32.0) | 84.1 (34.9)

2. Secondary Outcome: Incidence of Efficacy Failure
Description: Efficacy failure was defined as the composite endpoint of biopsy-proven acute rejection (BPAR), graft loss, death, lost to follow-up (from any reason), whichever occurred first. Incidence of efficacy failure was estimated using crude rate estimation (relative frequency).
Time Frame: Month 11
Population: ITT
Measure: Number; unit: Percentage of participants
Arm/Group | Everolimus | Calcineurin Inhibitor (CNI)
Number analyzed (Participants) | 96 | 98
Percentage of participants | 20.8 | 20.4

3. Secondary Outcome: Incidence of the Need for a Change in the Immunosuppressive Regimen
Description: The incidence of any changes in the immunosuppressive regimen other than allowed in the study protocol (for example, introduction of Mycophenolic acid (MPA) or sirolimus) was estimated using crude rate estimation (relative frequency).
Time Frame: Month 11
Population: ITT
Measure: Number; unit: Percentage of participants
Arm/Group | Everolimus | Calcineurin Inhibitor (CNI)
Number analyzed (Participants) | 96 | 98
Percentage of participants | 80.2 | 73.5

4. Secondary Outcome: Incidence of Renal Deterioration
Description: Renal deterioration was defined as a decrease by ≥25% in the cGFR compared to baseline and confirmed by one consecutive measurement. The analysis of this outcome measure was omitted because of missing relevance.
Time Frame: Baseline, Month 11
Reporting Status: Not Posted

5. Secondary Outcome: Renal Function (cGFR)
Description: This outcome measure evaluated renal function by assessing the calculated GFR based on the Cockcroft-Gault formula.
Time Frame: Month 5
Population: ITT
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Everolimus | Calcineurin Inhibitor (CNI)
Number analyzed (Participants) | 96 | 98
mL/min | 88.7 (31.0) | 82.9 (29.4)

6. Secondary Outcome: Incidence of Treated BPAR
Description: The incidence of treated BPAR was estimated using crude rate estimation (relative frequency).
Time Frame: Month 11
Population: ITT
Measure: Number; unit: Percentage of Participants
Arm/Group | Everolimus | Calcineurin Inhibitor (CNI)
Number analyzed (Participants) | 96 | 98
Percentage of Participants | 13.5 | 10.2

7. Secondary Outcome: Patient and Graft Survival
Description: Patient survival was defined as the time from date of randomization to date of death from any cause. If a patient was not known to have died, patient survival was censored as the date of last contact. Graft survival was defined as the time from the date of randomization to the date of graft loss. If a patient was not known to suffer from a graft loss or died without graft loss, time to graft loss was censored with date of last contact or date of death, respectively. Patient and graft survival were analyzed using the Kaplan Meier method.
Time Frame: Month 11
Population: ITT
Measure: Number; unit: Percentage of Participants
Arm/Group | Everolimus | Calcineurin Inhibitor (CNI)
Number analyzed (Participants) | 96 | 98
Percentage of Participants
  Death | 4.3 | 4.1
  Graft loss | 2.2 | 2.1

8. Secondary Outcome: Hepatitis C Virus (HCV) Replication in HCV-positive Patients
Description: HCV ribonucleic acid (RNA) was measured by real time reverse transcriptase polymerase chain reaction (PCR; copies per mL).
Time Frame: Baseline, Month 5
Population: ITT
Measure: Number; unit: Percentage of participants
Arm/Group | Everolimus | Calcineurin Inhibitor (CNI)
Number analyzed (Participants) | 96 | 98
Percentage of participants
  Baseline, negative | 64.5 | 55.3
  Baseline, positive | 0.0 | 0.0
  Baseline, not done | 35.5 | 44.7
  Month 5, negative | 62.9 | 38.2
  Month 5, positive | 1.6 | 13.2
  Month 5, not done | 35.5 | 48.7

9. Secondary Outcome: Number of Patients Who Experienced Adverse Events, Serious Adverse Events and Death
Description: Patients with all (serious and non-serious) adverse events, serious adverse events and death were reported.
Time Frame: From randomization to Month 11
Population: Safety population: This set included all randomized patients with at least one post-baseline measurement of GFR.
Measure: Number; unit: Number of participants
Arm/Group | Everolimus | Calcineurin Inhibitor (CNI)
Number analyzed (Participants) | 101 | 102
Number of participants
  Adverse Events (serious and non-serious) | 98 | 96
  Serious Adverse Events | 67 | 58
  Deaths | 4 | 4

10. Secondary Outcome: Number of Patients Who Experienced Adverse Events, Serious Adverse Events and Death
Description: Patients with all (serious and non-serious) adverse events, serious adverse events and death were reported.
Time Frame: Month 12 to Month 59 post-baseline
Population: Safety population: This set included all randomized patients with at least one post-baseline measurement of GFR.
Measure: Number; unit: Number of participants
Arm/Group | Everolimus | Calcineurin Inhibitor (CNI)
Number analyzed (Participants) | 41 | 40
Number of participants
  Adverse Events (serious and non-serious) | 41 | 40
  Serious Adverse Events | 26 | 28
  Deaths | 1 | 2

ADVERSE EVENTS:
Groups:
- Extension Period - Everolimus: Basiliximab plus everolimus-based immunosuppressive regimen following the reduction and cessation of initial CNI regimen plus optional steroids according to local best practice
- Extension Period - CNI: Basiliximab plus CNI-based immunosuppressive regimen according to local best practice plus optional steroids according to local best practice
Arm/Group | Everolimus | Calcineurin Inhibitor (CNI) | Extension Period - Everolimus | Extension Period - CNI
Serious Adverse Events (participants affected / at risk) | 67/101 | 58/102 | 26/41 | 28/40
Other Adverse Events (participants affected / at risk) | 92/101 | 87/102 | 39/41 | 38/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus (N=101) | Calcineurin Inhibitor (CNI) (N=102) | Extension Period - Everolimus (N=41) | Extension Period - CNI (N=40)
ANAEMIA (Blood and lymphatic system disorders) | 3 | 2 | 0 | 1
DISSEMINATED INTRAVASCULAR COAGULATION (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
HAEMOLYTIC URAEMIC SYNDROME (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
LEUKOPENIA (Blood and lymphatic system disorders) | 4 | 0 | 0 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
PANCYTOPENIA (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
THROMBOTIC MICROANGIOPATHY (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 0 | 0 | 1
ARRHYTHMIA (Cardiac disorders) | 1 | 0 | 0 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 0 | 1 | 0
ATRIOVENTRICULAR BLOCK (Cardiac disorders) | 1 | 0 | 0 | 0
BUNDLE BRANCH BLOCK RIGHT (Cardiac disorders) | 0 | 0 | 1 | 0
CARDIAC ARREST (Cardiac disorders) | 0 | 1 | 0 | 0
CARDIAC FAILURE (Cardiac disorders) | 1 | 0 | 0 | 0
CARDIAC FAILURE ACUTE (Cardiac disorders) | 0 | 1 | 0 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 1 | 0 | 0
PERICARDIAL EFFUSION (Cardiac disorders) | 2 | 0 | 0 | 0
TACHYCARDIA (Cardiac disorders) | 1 | 0 | 0 | 0
TORSADE DE POINTES (Cardiac disorders) | 1 | 0 | 0 | 0
VERTIGO (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
GOITRE (Endocrine disorders) | 1 | 0 | 0 | 1
HYPERTHYROIDISM (Endocrine disorders) | 1 | 0 | 0 | 0
TOXIC NODULAR GOITRE (Endocrine disorders) | 1 | 0 | 0 | 0
MACULAR OEDEMA (Eye disorders) | 1 | 0 | 0 | 0
OCULAR ICTERUS (Eye disorders) | 1 | 0 | 0 | 0
PAPILLOEDEMA (Eye disorders) | 1 | 0 | 0 | 0
RETINAL HAEMORRHAGE (Eye disorders) | 1 | 0 | 0 | 0
RETINAL VEIN OCCLUSION (Eye disorders) | 0 | 1 | 0 | 0
RETINITIS (Eye disorders) | 0 | 1 | 0 | 0
ABDOMINAL HERNIA (Gastrointestinal disorders) | 0 | 0 | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 4 | 2 | 0 | 0
ANAL PROLAPSE (Gastrointestinal disorders) | 0 | 1 | 0 | 0
ASCITES (Gastrointestinal disorders) | 0 | 2 | 1 | 1
COELIAC ARTERY STENOSIS (Gastrointestinal disorders) | 0 | 1 | 0 | 0
CROHN'S DISEASE (Gastrointestinal disorders) | 0 | 0 | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 1 | 1 | 0 | 0
DYSPHAGIA (Gastrointestinal disorders) | 0 | 0 | 0 | 1
GASTRITIS (Gastrointestinal disorders) | 0 | 1 | 0 | 0
GASTRITIS HAEMORRHAGIC (Gastrointestinal disorders) | 0 | 1 | 0 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 1 | 0 | 0
GASTROINTESTINAL NECROSIS (Gastrointestinal disorders) | 0 | 0 | 1 | 0
ILEUS (Gastrointestinal disorders) | 0 | 2 | 1 | 0
ILEUS PARALYTIC (Gastrointestinal disorders) | 0 | 0 | 0 | 1
INGUINAL HERNIA (Gastrointestinal disorders) | 2 | 1 | 1 | 0
INTESTINAL DILATATION (Gastrointestinal disorders) | 0 | 1 | 0 | 0
INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1 | 0 | 0
MALABSORPTION (Gastrointestinal disorders) | 0 | 0 | 1 | 0
MECHANICAL ILEUS (Gastrointestinal disorders) | 0 | 1 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 1 | 2 | 0 | 1
OESOPHAGEAL VARICES HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 0 | 1
PANCREATIC CYST (Gastrointestinal disorders) | 0 | 1 | 0 | 0
PANCREATITIS (Gastrointestinal disorders) | 0 | 3 | 0 | 0
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 | 0 | 1 | 0
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 1 | 0 | 0
SMALL INTESTINAL STENOSIS (Gastrointestinal disorders) | 0 | 1 | 0 | 0
SUBILEUS (Gastrointestinal disorders) | 1 | 0 | 0 | 0
UMBILICAL HERNIA (Gastrointestinal disorders) | 0 | 0 | 1 | 0
VOMITING (Gastrointestinal disorders) | 2 | 1 | 0 | 2
ASTHENIA (General disorders) | 0 | 1 | 0 | 0
CHEST PAIN (General disorders) | 1 | 0 | 0 | 0
CONCOMITANT DISEASE PROGRESSION (General disorders) | 1 | 0 | 0 | 0
CYST (General disorders) | 0 | 0 | 0 | 1
DEATH (General disorders) | 1 | 0 | 0 | 0
DISEASE PROGRESSION (General disorders) | 3 | 0 | 0 | 0
DRUG INEFFECTIVE (General disorders) | 2 | 0 | 0 | 0
DRUG INTERACTION (General disorders) | 0 | 0 | 0 | 1
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 1 | 0 | 0 | 0
HERNIA (General disorders) | 1 | 0 | 0 | 0
HERNIA PAIN (General disorders) | 0 | 1 | 0 | 0
INFLAMMATION (General disorders) | 1 | 0 | 0 | 0
MULTI-ORGAN FAILURE (General disorders) | 0 | 1 | 0 | 0
OEDEMA PERIPHERAL (General disorders) | 1 | 0 | 0 | 0
PYREXIA (General disorders) | 6 | 4 | 2 | 1
BILE DUCT OBSTRUCTION (Hepatobiliary disorders) | 0 | 1 | 0 | 0
BILE DUCT STENOSIS (Hepatobiliary disorders) | 2 | 5 | 1 | 2
BILIARY ISCHAEMIA (Hepatobiliary disorders) | 2 | 4 | 2 | 2
BILIARY TRACT DISORDER (Hepatobiliary disorders) | 1 | 0 | 0 | 0
BILOMA (Hepatobiliary disorders) | 1 | 0 | 0 | 0
CHOLANGITIS (Hepatobiliary disorders) | 4 | 10 | 1 | 3
CHOLELITHIASIS (Hepatobiliary disorders) | 0 | 1 | 0 | 0
CHOLESTASIS (Hepatobiliary disorders) | 5 | 2 | 0 | 0
HEPATIC ARTERY OCCLUSION (Hepatobiliary disorders) | 0 | 0 | 0 | 1
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 0 | 0 | 0 | 1
HEPATIC FAILURE (Hepatobiliary disorders) | 0 | 0 | 0 | 1
HEPATIC HAEMORRHAGE (Hepatobiliary disorders) | 0 | 1 | 0 | 0
HEPATIC LESION (Hepatobiliary disorders) | 0 | 0 | 0 | 1
HEPATIC STEATOSIS (Hepatobiliary disorders) | 1 | 0 | 0 | 1
HEPATIC VEIN THROMBOSIS (Hepatobiliary disorders) | 0 | 0 | 1 | 0
HEPATITIS (Hepatobiliary disorders) | 0 | 1 | 0 | 0
HEPATORENAL SYNDROME (Hepatobiliary disorders) | 0 | 0 | 0 | 1
HEPATOTOXICITY (Hepatobiliary disorders) | 2 | 1 | 0 | 0
NON-ALCOHOLIC STEATOHEPATITIS (Hepatobiliary disorders) | 0 | 0 | 1 | 0
PORTAL VEIN THROMBOSIS (Hepatobiliary disorders) | 0 | 0 | 1 | 0
HYPERSENSITIVITY (Immune system disorders) | 0 | 1 | 0 | 0
LIVER TRANSPLANT REJECTION (Immune system disorders) | 4 | 1 | 0 | 0
TRANSPLANT REJECTION (Immune system disorders) | 1 | 1 | 0 | 0
ABDOMINAL ABSCESS (Infections and infestations) | 1 | 1 | 0 | 0
ASPERGILLOSIS (Infections and infestations) | 0 | 0 | 0 | 1
BILIARY SEPSIS (Infections and infestations) | 0 | 1 | 0 | 0
BRAIN ABSCESS (Infections and infestations) | 1 | 0 | 0 | 0
BRONCHITIS (Infections and infestations) | 0 | 0 | 0 | 1
BRONCHOPNEUMONIA (Infections and infestations) | 0 | 1 | 0 | 1
BRONCHOPULMONARY ASPERGILLOSIS (Infections and infestations) | 0 | 1 | 0 | 0
CELLULITIS (Infections and infestations) | 1 | 0 | 0 | 0
CELLULITIS ORBITAL (Infections and infestations) | 0 | 0 | 1 | 0
CEREBRAL TOXOPLASMOSIS (Infections and infestations) | 1 | 0 | 0 | 0
CLOSTRIDIAL INFECTION (Infections and infestations) | 1 | 0 | 0 | 0
CLOSTRIDIUM COLITIS (Infections and infestations) | 0 | 0 | 1 | 0
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 1 | 0 | 0 | 0
CYTOMEGALOVIRUS COLITIS (Infections and infestations) | 1 | 0 | 0 | 0
CYTOMEGALOVIRUS INFECTION (Infections and infestations) | 1 | 5 | 1 | 0
DEVICE RELATED INFECTION (Infections and infestations) | 1 | 0 | 0 | 0
DIVERTICULITIS (Infections and infestations) | 1 | 0 | 1 | 0
ENDOCARDITIS (Infections and infestations) | 1 | 0 | 1 | 0
ENTEROCOCCAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 1
ENTEROCOCCAL SEPSIS (Infections and infestations) | 0 | 1 | 0 | 0
ERYSIPELAS (Infections and infestations) | 0 | 1 | 0 | 0
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 0 | 1 | 0 | 0
GASTROENTERITIS (Infections and infestations) | 0 | 1 | 1 | 2
GASTROENTERITIS NOROVIRUS (Infections and infestations) | 1 | 0 | 0 | 0
GASTROINTESTINAL INFECTION (Infections and infestations) | 0 | 1 | 0 | 1
HAEMATOMA INFECTION (Infections and infestations) | 0 | 0 | 0 | 1
HEPATITIS C (Infections and infestations) | 3 | 3 | 0 | 1
HERPES ZOSTER (Infections and infestations) | 0 | 0 | 0 | 1
INCISIONAL HERNIA GANGRENOUS (Infections and infestations) | 0 | 1 | 0 | 0
INFECTION (Infections and infestations) | 1 | 0 | 2 | 2
LIVER ABSCESS (Infections and infestations) | 3 | 0 | 0 | 0
OESOPHAGEAL CANDIDIASIS (Infections and infestations) | 0 | 0 | 0 | 1
PANCREATITIS BACTERIAL (Infections and infestations) | 0 | 1 | 0 | 0
PERIHEPATIC ABSCESS (Infections and infestations) | 0 | 1 | 0 | 0
PERITONEAL ABSCESS (Infections and infestations) | 0 | 1 | 0 | 0
PERITONITIS BACTERIAL (Infections and infestations) | 0 | 1 | 0 | 1
PNEUMOCYSTIS JIROVECI PNEUMONIA (Infections and infestations) | 1 | 0 | 0 | 0
PNEUMONIA (Infections and infestations) | 5 | 3 | 1 | 2
PNEUMONIA CYTOMEGALOVIRAL (Infections and infestations) | 1 | 0 | 1 | 0
PNEUMONIA PRIMARY ATYPICAL (Infections and infestations) | 0 | 1 | 0 | 0
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0 | 1 | 0
SEPSIS (Infections and infestations) | 2 | 2 | 1 | 0
SEPTIC SHOCK (Infections and infestations) | 0 | 0 | 0 | 1
SMALL INTESTINE GANGRENE (Infections and infestations) | 0 | 1 | 0 | 0
STENOTROPHOMONAS INFECTION (Infections and infestations) | 0 | 0 | 0 | 1
TONSILLITIS (Infections and infestations) | 1 | 0 | 0 | 0
URINARY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0 | 1
WOUND INFECTION (Infections and infestations) | 1 | 0 | 0 | 0
ANASTOMOTIC STENOSIS (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 0
ANIMAL BITE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
BILIARY ANASTOMOSIS COMPLICATION (Injury, poisoning and procedural complications) | 4 | 3 | 0 | 0
FALL (Injury, poisoning and procedural complications) | 1 | 1 | 3 | 1
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
FOOT FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 8 | 5 | 7 | 5
INCISIONAL HERNIA, OBSTRUCTIVE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
LIVER GRAFT LOSS (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 0
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0
PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
RIB FRACTURE (Injury, poisoning and procedural complications) | 2 | 0 | 2 | 0
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0
TRANSPLANT FAILURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
WOUND COMPLICATION (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
WRIST FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0 | 0 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0 | 0 | 0
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 1 | 0 | 0 | 0
BLOOD CREATININE INCREASED (Investigations) | 0 | 0 | 0 | 1
C-REACTIVE PROTEIN INCREASED (Investigations) | 2 | 1 | 0 | 1
CYTOMEGALOVIRUS TEST POSITIVE (Investigations) | 1 | 0 | 0 | 0
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 2 | 0 | 0 | 0
HAEMOGLOBIN DECREASED (Investigations) | 0 | 1 | 0 | 0
HEPATIC ENZYME INCREASED (Investigations) | 14 | 9 | 1 | 1
LIVER FUNCTION TEST ABNORMAL (Investigations) | 3 | 1 | 0 | 0
TRANSAMINASES INCREASED (Investigations) | 4 | 3 | 1 | 1
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
ELECTROLYTE IMBALANCE (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 | 3 | 0 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
HYPOVITAMINOSIS (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
OSTEOPENIA (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
OSTEOPOROTIC FRACTURE (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
BLADDER TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
EPSTEIN-BARR VIRUS ASSOCIATED LYMPHOPROLIFERATIVE DISORDER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
HEPATIC NEOPLASM MALIGNANT RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
HEPATOCELLULAR CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 1
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
METASTASES TO BONE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
METASTASES TO LUNG (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
METASTASES TO LYMPH NODES (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
METASTASES TO PERITONEUM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
PARANEOPLASTIC SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
PROSTATE CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
RECTAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
APHASIA (Nervous system disorders) | 1 | 0 | 0 | 0
CAROTID ARTERY STENOSIS (Nervous system disorders) | 0 | 0 | 0 | 1
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 0 | 0 | 0 | 1
CEREBRAL INFARCTION (Nervous system disorders) | 1 | 0 | 1 | 0
CEREBRAL ISCHAEMIA (Nervous system disorders) | 0 | 0 | 0 | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 0 | 0 | 1
DIZZINESS (Nervous system disorders) | 1 | 0 | 0 | 0
ENCEPHALOPATHY (Nervous system disorders) | 1 | 0 | 0 | 0
EPILEPSY (Nervous system disorders) | 1 | 0 | 0 | 0
GRAND MAL CONVULSION (Nervous system disorders) | 0 | 1 | 0 | 0
HEMIPARESIS (Nervous system disorders) | 0 | 0 | 0 | 1
LACUNAR INFARCTION (Nervous system disorders) | 0 | 0 | 0 | 1
LETHARGY (Nervous system disorders) | 0 | 1 | 0 | 0
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 1 | 0 | 0 | 0
MIGRAINE (Nervous system disorders) | 1 | 0 | 0 | 0
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 | 0 | 0 | 0
NEUROTOXICITY (Nervous system disorders) | 0 | 1 | 0 | 0
PARAESTHESIA (Nervous system disorders) | 1 | 0 | 0 | 0
POLYNEUROPATHY (Nervous system disorders) | 0 | 0 | 1 | 0
RADICULAR SYNDROME (Nervous system disorders) | 0 | 0 | 0 | 1
SOMNOLENCE (Nervous system disorders) | 0 | 1 | 0 | 1
SYNCOPE (Nervous system disorders) | 0 | 1 | 0 | 1
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 | 1 | 0 | 1
ALCOHOLISM (Psychiatric disorders) | 0 | 0 | 1 | 0
DEPRESSION (Psychiatric disorders) | 1 | 0 | 0 | 0
DISORIENTATION (Psychiatric disorders) | 0 | 1 | 0 | 0
PSYCHOTIC DISORDER DUE TO A GENERAL MEDICAL CONDITION (Psychiatric disorders) | 0 | 0 | 0 | 1
SUICIDE ATTEMPT (Psychiatric disorders) | 0 | 1 | 0 | 1
HAEMATURIA (Renal and urinary disorders) | 1 | 0 | 0 | 0
RENAL FAILURE (Renal and urinary disorders) | 0 | 1 | 0 | 0
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 | 0 | 1 | 0
RENAL IMPAIRMENT (Renal and urinary disorders) | 0 | 1 | 0 | 0
RENAL INJURY (Renal and urinary disorders) | 0 | 0 | 0 | 1
MENORRHAGIA (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
OVARIAN CYST (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
SPERMATOCELE (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
TESTICULAR SWELLING (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
LUNG INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 1
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
VOCAL CORD POLYP (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
SCAR (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
TOXIC SKIN ERUPTION (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
CIRCULATORY COLLAPSE (Vascular disorders) | 0 | 1 | 1 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 0 | 1 | 0
HYPERTENSIVE CRISIS (Vascular disorders) | 1 | 1 | 0 | 1
SHOCK HAEMORRHAGIC (Vascular disorders) | 1 | 0 | 0 | 0
STEAL SYNDROME (Vascular disorders) | 1 | 0 | 0 | 0
VENA CAVA THROMBOSIS (Vascular disorders) | 0 | 1 | 0 | 0
VENOUS STENOSIS (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus (N=101) | Calcineurin Inhibitor (CNI) (N=102) | Extension Period - Everolimus (N=41) | Extension Period - CNI (N=40)
ANAEMIA (Blood and lymphatic system disorders) | 17 | 10 | 4 | 1
LEUKOPENIA (Blood and lymphatic system disorders) | 19 | 10 | 1 | 3
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 8 | 7 | 2 | 4
TACHYCARDIA (Cardiac disorders) | 6 | 2 | 0 | 0
HYPOTHYROIDISM (Endocrine disorders) | 0 | 0 | 1 | 2
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 2 | 1 | 0 | 2
ABDOMINAL PAIN (Gastrointestinal disorders) | 11 | 10 | 4 | 2
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 6 | 6 | 5 | 2
APHTHOUS STOMATITIS (Gastrointestinal disorders) | 8 | 1 | 2 | 0
ASCITES (Gastrointestinal disorders) | 1 | 8 | 1 | 2
CONSTIPATION (Gastrointestinal disorders) | 9 | 11 | 1 | 3
DIARRHOEA (Gastrointestinal disorders) | 27 | 13 | 10 | 4
FLATULENCE (Gastrointestinal disorders) | 7 | 10 | 5 | 2
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 2 | 1 | 4 | 2
NAUSEA (Gastrointestinal disorders) | 12 | 16 | 5 | 3
VOMITING (Gastrointestinal disorders) | 6 | 12 | 3 | 0
FATIGUE (General disorders) | 5 | 6 | 2 | 3
IMPAIRED HEALING (General disorders) | 0 | 1 | 2 | 2
OEDEMA (General disorders) | 5 | 6 | 0 | 0
OEDEMA PERIPHERAL (General disorders) | 15 | 9 | 13 | 3
PYREXIA (General disorders) | 14 | 12 | 4 | 3
CHOLANGITIS (Hepatobiliary disorders) | 6 | 5 | 1 | 1
CHOLESTASIS (Hepatobiliary disorders) | 9 | 4 | 2 | 1
HEPATIC STEATOSIS (Hepatobiliary disorders) | 2 | 4 | 6 | 5
BRONCHITIS (Infections and infestations) | 2 | 1 | 6 | 6
CYTOMEGALOVIRUS INFECTION (Infections and infestations) | 7 | 7 | 1 | 0
NASOPHARYNGITIS (Infections and infestations) | 15 | 15 | 9 | 8
PERIODONTITIS (Infections and infestations) | 0 | 0 | 5 | 2
SINUSITIS (Infections and infestations) | 6 | 1 | 4 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 2 | 4 | 1
URINARY TRACT INFECTION (Infections and infestations) | 16 | 13 | 6 | 4
WOUND INFECTION (Infections and infestations) | 7 | 2 | 2 | 0
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 4 | 5 | 7 | 2
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 4 | 8 | 3 | 1
C-REACTIVE PROTEIN INCREASED (Investigations) | 8 | 2 | 2 | 1
HEPATIC ENZYME INCREASED (Investigations) | 14 | 3 | 0 | 4
TRANSAMINASES INCREASED (Investigations) | 8 | 6 | 4 | 1
WEIGHT DECREASED (Investigations) | 1 | 1 | 1 | 2
DIABETES MELLITUS (Metabolism and nutrition disorders) | 4 | 6 | 5 | 2
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 22 | 11 | 4 | 2
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 | 7 | 0 | 2
HYPERLIPIDAEMIA (Metabolism and nutrition disorders) | 12 | 2 | 1 | 0
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 6 | 3 | 2 | 1
HYPERURICAEMIA (Metabolism and nutrition disorders) | 5 | 7 | 2 | 3
HYPOKALAEMIA (Metabolism and nutrition disorders) | 13 | 9 | 3 | 1
OBESITY (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 7 | 10 | 3 | 2
BACK PAIN (Musculoskeletal and connective tissue disorders) | 12 | 13 | 9 | 1
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 4 | 7 | 1 | 1
OSTEOPENIA (Musculoskeletal and connective tissue disorders) | 0 | 3 | 2 | 2
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 2 | 4 | 6 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 5 | 6 | 7 | 0
MELANOCYTIC NAEVUS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 2
HEADACHE (Nervous system disorders) | 20 | 10 | 3 | 1
PARAESTHESIA (Nervous system disorders) | 4 | 4 | 3 | 1
TREMOR (Nervous system disorders) | 6 | 9 | 0 | 0
DEPRESSION (Psychiatric disorders) | 3 | 6 | 2 | 7
INSOMNIA (Psychiatric disorders) | 8 | 9 | 1 | 2
SLEEP DISORDER (Psychiatric disorders) | 4 | 6 | 4 | 1
PROTEINURIA (Renal and urinary disorders) | 10 | 2 | 4 | 0
RENAL FAILURE (Renal and urinary disorders) | 3 | 7 | 2 | 6
RENAL FAILURE CHRONIC (Renal and urinary disorders) | 0 | 2 | 0 | 2
URINARY INCONTINENCE (Renal and urinary disorders) | 0 | 0 | 0 | 2
METRORRHAGIA (Reproductive system and breast disorders) | 1 | 0 | 0 | 2
COUGH (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 4 | 2
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 0 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 9 | 8 | 1 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 19 | 11 | 5 | 4
RASH (Skin and subcutaneous tissue disorders) | 5 | 1 | 1 | 3
HYPERTENSION (Vascular disorders) | 20 | 14 | 6 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.